CLINICAL TRIAL: NCT00715689
Title: Dose Study Investigating Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of NNC126-0083 in Growth Hormone Deficient Adults (GHDA)
Brief Title: Dose Study in Growth Hormone Deficient Adults Investigating Safety, Pharmacokinetics and Pharmacodynamics of NNC126-0083
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8630-1823; 2008-001061-29 (EudraCT Number)
Record Dates: First submitted 2008-07-14; First posted 2008-07-15 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Growth Hormone Disorder; Adult Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — NNC126-0083

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental)
  Interventions: Drug: NNC126-0083; Drug: placebo
- B (Experimental)
  Interventions: Drug: NNC126-0083; Drug: placebo
- C (Experimental)
  Interventions: Drug: NNC126-0083; Drug: placebo
- D (Experimental)
  Interventions: Drug: NNC126-0083; Drug: placebo

INTERVENTIONS:
Drug: NNC126-0083 — Dose level 1; (6 subjects active, 2 subjects placebo); s.c. injection once weekly for 3 weeks
  Other Names: pegylated long-acting human growth hormone
  Arms: A
Drug: NNC126-0083 — Dose level 2; (6 subjects active, 2 subjects placebo); s.c. injection once weekly for 3 weeks
  Other Names: pegylated long-acting human growth hormone
  Arms: B
Drug: NNC126-0083 — Dose level 3; (6 subjects active, 2 subjects placebo); s.c. injection once weekly for 3 weeks
  Other Names: pegylated long-acting human growth hormone
  Arms: C
Drug: NNC126-0083 — Dose level 4; (6 subjects active, 2 subjects placebo); s.c. injection once weekly for 3 weeks
  Other Names: pegylated long-acting human growth hormone
  Arms: D
Drug: placebo — Dose level 1; NNC126-0083 placebo for s.c. injection once weekly for 3 weeks
  Arms: A
Drug: placebo — Dose level 2; NNC126-0083 placebo for s.c. injection once weekly for 3 weeks
  Arms: B
Drug: placebo — Dose level 3; NNC126-0083 placebo for s.c. injection once weekly for 3 weeks
  Arms: C
Drug: placebo — Dose level 4; NNC126-0083 placebo for s.c. injection once weekly for 3 weeks
  Arms: D

SUMMARY:
This trial is conducted in Europe. The aim of this clinical trial is to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of NNC126-0083 in growth hormone deficient adults

ELIGIBILITY:
Inclusion Criteria:

* GHDA subjects as defined in the Consensus guidelines for the diagnosis and treatment of adults with GH deficiency II
* Fertile females must agree to use appropriate contraceptive methods and have a negative pregnancy test at inclusion
* GH replacement therapy for more than 3 months
* Body Mass Index (BMI, kg/m2) of 22.0 to 35.0 kg/m2, both inclusive

Exclusion Criteria:

* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods
* Malignant disease
* Proliferative retinopathy judged by retina-photo within the last year - only with concomitant diabetes
* Heart insufficiency, NYHA class greater than 2
* Subjects with diabetes with an HbA1C above 8.0%
* Diabetic receiving insulin treatment
* Stable pituitary replacement therapy for less than 3 months
* Impaired liver function
* Impaired kidney function

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (adverse events, local tolerability, physical examination) | 0 to 10 days after third dosing, (day 15-25 after first dose)

SECONDARY OUTCOMES:
Cmax, maximum concentration of IGF-I | after trial product administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (3):
- Denmark (3):
  - Novo Nordisk Investigational Site, Århus C
  - Novo Nordisk Investigational Site, København Ø
  - Novo Nordisk Investigational Site, Odense

REFERENCES:
- [Result] Sondergaard E, Klose M, Hansen M, Hansen BS, Andersen M, Feldt-Rasmussen U, Laursen T, Rasmussen MH, Christiansen JS. Pegylated long-acting human growth hormone possesses a promising once-weekly treatment profile, and multiple dosing is well tolerated in adult patients with growth hormone deficiency. J Clin Endocrinol Metab. 2011 Mar;96(3):681-8. doi: 10.1210/jc.2010-1931. Epub 2010 Dec 22. PMID 21177789
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com